CLINICAL TRIAL: NCT03148132
Title: Comparison of the Vascular Endothelial Growth Factor Serum Concentrations After Intravitreal Use of Bevacizumab or Ranibizumab as a Treatment for Type 1 Retinopathy of Prematurity
Brief Title: VEGF Concentrations After Intravitreal Bevacizumab vs Ranibizumab as a Treatment for Type 1 ROP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidad Autonoma de San Luis Potosí (Other)
Collaborators: Hospital Central "Dr. Ignacio Morones Prieto" (Other)
Responsible Party: Principal Investigator, Ada Gabriela Hernández Gámez, MD, Universidad Autonoma de San Luis Potosí
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 31-17
Record Dates: First submitted 2017-05-08; First posted 2017-05-10 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Retinopathy of Prematurity Both Eyes; Retinal Disease; Premature Birth; Eye Diseases
Keywords: Retinopathy of Prematurity; VEGF; Bevacizumab; Ranibizumab
MeSH Terms: conditions — Retinal Diseases; Premature Birth; Eye Diseases; Retinopathy of Prematurity | interventions — Bevacizumab; Intravitreal Injections

STUDY DESIGN:
Intervention Model Description: Group 1: Patients that fullfil type 1 ROP criteria that will be treated with Bevacizumab Group 2: Patients that fullfil type 1 ROP criteria that will be treated with Ranibizumab
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The principal investigator and the outcomes assesor will be blinded, the assignation of the treatment will be randomized. The parents or tutor of the participant will be blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bevacizumab injection (Active Comparator): Application of Intravitreal Bevacizumab (0.50mg/0.02mL), unique dosis
  Interventions: Drug: Bevacizumab Injection
- Ranibizumab Ophthalmic (Experimental): Application of Intravitreal Ranibizumab (0.25mg/0.025mL), unique dosis
  Interventions: Drug: Ranibizumab Ophthalmic

INTERVENTIONS:
Drug: Bevacizumab Injection — 0.5mg/0.02 mL
  Other Names: Intravitreal
  Arms: Bevacizumab injection
Drug: Ranibizumab Ophthalmic — 0.25mg/0.025 mL
  Other Names: Intravitreal
  Arms: Ranibizumab Ophthalmic

SUMMARY:
The Retinopathy of Prematurity (ROP) is one of the leading causes of blindness on the pediatric age worldwide. This pathology is characterized for arrest of the normal vascular and neuronal retina that because of pathological compensatory mechanisms results in proliferation of vascular tissue that grow in the limit between the vascular retina and the avascular retina.

The ET-ROP group classified the ROP by those who need treatment immediately or those who doesn't need treatment, The classification is the following Type 1 ROP-->ROP zone I any stage with plus, zone I stage 3 without plus, zone II stage 2 y 3 with plus Type 2 ROP --> Zone 1, Stage 2 or 3 without plus, and Zone II, stage 3 without plus.

The treatment is begun on patient with type 1 ROP and type 2 ROP is maintained in observation.

DETAILED DESCRIPTION:
It has been documented that de Vascular Endothelial Growth Factor (VEGF) is involved on the physiopathology of this disease.

The VEGF is a glucoprotein that regulates the angiogenesis and the vasculogenesis, it's presence is crucial on the growth and development of several tissues around the organism.

Nowadays the treatment of type 1 ROP it si focus on the disminution of the intravitreal VEGF after the intravitreal application of drugs like Bevacizumab and Ranibizumab.

However these drugs can pass through the hematorretinal barrier in to the blood stream where they can also decrease the systemic levels of VEGF.

We still don't know the long term effects of the intravitreal application of these drugs on premature babies, but there is the concern.

The objective of this study is to compare the serum VEGF concentrations after intravitreal application of Bevacizumab (0.500mg/0.02mL) versus Ranibizumab (0.25 mg/0.025mL) for the treatment of type 1 ROP.

HYPOTESIS: The serum VEGF concentrations after the intravitreal application of Bevacizumab will be smaller than the serum VEGF concentrations after the intravitreal application of Ranibizumab.

METHODOLOGY: Safety ECCA. Inclusion criteria, premature newborns who fulfill the criteria for type 1 ROP according to the ET-ROP classification.

The investigators will identify the patients that can be included The principal investigator will take a blood sample of 500 microliters and then the patients would receive intravitreal treatment assigned randomly (Bevacizumab 0.5mg/0.02mL or Ranibizumab 0.25mg/0.25 mL).

The principal investigator will take new blood samples a day, 2 weeks and 8 weeks after the application of the intravitreal treatment, these samples will be frozen to further analysis.

The analysis will be performed by ELISA kits.

The investigators are going to describe the results of the ELISA for the blood samples, and then make a comparison between both groups.

ELIGIBILITY:
Inclusion Criteria:

* Premature newborns that fulfill the criteria for type 1 ROP, according to the Early Treatment of ROP classification on both eyes.

Exclusion Criteria:

* Patients that do not continue the required evaluations.

Ages: 28 Days to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2017-05-23 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
To compare the serum VEGF concentrations after intravitreal application of Bevacizumab vs Ranibizumab | 6 months
  Evaluate the Serum VEGF concentration with the ELISA assay after intravitreal application of Bevacizumab or ranibizumab

CONTACTS AND LOCATIONS:
Overall Officials: Martha G Rangel, MD, Study Director — Hospital Central "Dr. Ignacio Morones Prieto"
Locations (1):
- Hospital Central "Dr. Ignacio Morones Prieto", San Luis Potosí City, Mexico

IPD SHARING:
Plan to Share IPD: No